CLINICAL TRIAL: NCT04981353
Title: Thoracic Erector Spinae Plane Block for painless1st Stage Normal Vaginal Delivery: Randomized Controlled Study
Brief Title: Thoracic Erector Spinae Plane Block for Painless 1st Stage Normal Vaginal Delivery: Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa adel, lecturer of anesthesia and intensive care MD, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU R 134/2021
Record Dates: First submitted 2021-07-23; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Numerical Rating Pain Score; the Total Doses of Pethidine Needed Through-out Delivery Will be Measured; the Incidence of Failed Delivery and Need of Cesarean Section Will be Assessed; the Incidence of Transient Fetal Bradycardia or Deceleration After the Administration of the Block Will be Recorded; ABGAR Score of the Neonate
Keywords: erector spinae plane block, normal vaginal delivery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): :(group 1) will be putted in sitting position and disinfecting her back. A real-time high-frequency linear ultrasound will be used to do the thoracic (ESP) at the level of T11 by visualizing the transverse process of T11 thoracic vertebrae and erector spinae muscle and injecting a 20 ml of bupivacaine 0.25% bilaterally using an in-plane technique, a 20-gauge, 70-mm needle (Tuoren, Henan, China) will be advanced into the plane below (ESM) after injecting lidocaine 1% 2ml at the site of injection, Needle will be advanced with a cranial to caudal direction
  Interventions: Procedure: bilateral erector spinae plane block at T11
- group 2 (Active Comparator): (group 2) patients will receive pethidine 25mg doses if NRS >4.
  Interventions: Procedure: bilateral erector spinae plane block at T11

INTERVENTIONS:
Procedure: bilateral erector spinae plane block at T11 — A real-time high-frequency linear ultrasound will be used to do the thoracic (ESP) at the level of T11 by visualizing the transverse process of T11 thoracic vertebrae and erector spinae muscle and injecting a 20 ml of bupivacaine 0.25% bilaterally using an in-plane technique, a 20-gauge, 70-mm needle (Tuoren, Henan, China) will be advanced into the plane below (ESM) after injecting lidocaine 1% 2ml at the site of injection, Needle will be advanced with a cranial to caudal directio

SUMMARY:
this study will test a novel indication for bilateral erector spinae plane block (painless 1st stage normal vaginal delivery) it depends on the hypnosis that the erector spinae plane block blocks the visceral pain also by affecting the ventral rami, dorsal rami and rami communicants.

DETAILED DESCRIPTION:
Aim of the work In this article, the efficacy of bilateral thoracic (ESP) to provide painless delivery without affecting the motor power (walking painless labor) will be studded.

The main objective:

1. numerical rating pain score (NRS) during the course of delivery will be recorded and compared.

Other objectives:

1. the total doses of pethidine needed through-out delivery will be measured
2. the incidence of failed delivery and need of cesarean section will be assessed
3. the incidence of transient fetal bradycardia or deceleration after the administration of the block will be recorded
4. ABGAR score of the neonate immediately after delivery and after 5min, 10min,15min after delivery. Will be recorded

Inclusion criteria :

Pregnant ladies aged 20-40 years, ASA 2, either prime or multipara , 37-40 weeks of gestation scheduled for vaginal delivery will be included in the study Exclusion criteria Pregnant ladies with complicated pregnancy eg; IUGR, accidental hemorrhage, preeclampsia Pregnant ladies scheduled for cesarean section Place of work: Labor ward in obstetric Department, Ain Shams University Hospital.

Sample size: all patients legible for the study will be enrolled and randomly allocated into one of the two groups. sample size was calculated using PASS 11.0 and based on a study carried out by Boules,2020. Group sample size of 15 in group 1 and 15 in group 2 achieves 100% power to detect difference of -4.0 between the null hypothesis that both group means are 2.0 and the alternative hypothesis that the mean of group 2 is 6.0 with estimated group standard deviations of 0.3 and a significance level (alpha ) of 0.05000 using a two-sided two-sample t-test. Sample size was inflated by 20% to account for attrition problem.

Methodology :

After taking the approval from Ain shams university ethical committee and informed consent from the pregnant ladies that will be legible for the study, detailed medical history of the patient will be taken and patient will be transported to operating room and basic monitors including ( ECG, pulse oximetry, NIBP)will be attached and basic reading of CTG will be recorded after that patient will be enrolled in two groups :(group 1) will be putted in sitting position and disinfecting her back. A real-time high-frequency linear ultrasound will be used to do the thoracic (ESP) at the level of T11 by visualizing the transverse process of T11 thoracic vertebrae and erector spinae muscle and injecting a 20 ml of bupivacaine 0.25% bilaterally using an in-plane technique, a 20-gauge, 70-mm needle (Tuoren, Henan, China) will be advanced into the plane below (ESM) after injecting lidocaine 1% 2ml at the site of injection, Needle will be advanced with a cranial to caudal direction (Boules et al,2020). (group 2) patients will receive pethidine 25mg doses if NRS >4. Patients of both groups will be positioned semi setting and CTG will be attached to her , blood pressure and maternal pulsations will be recorded every 15min throughout the delivery process. CTG records all over the labor time will be printed. Numerical rating scale (NRS) are the simplest and most widely used scale. The numerical scale is most commonly 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable." The patient draws a circle around the number that best describes the pain intensity. Advantages of NRS include simplicity, reproducibility, easy comprehensibility, and sensitivity to small changes in pain. It will be assessed every 30 min. throughout the delivery process. 25mg pethidine iv will be given if NRS >4 in both groups.

Endpoints of this study:

One hour after delivery of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies 37-40 weeks of gestation scheduled for normal vaginal delivery ASA 2 either prime or multipara

Exclusion Criteria:

* pregnant ladies with complicated pregnancy eg; IUGR,accidental hemorrhage, preeclampsia pregnant ladies scheduled for cesarean section

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-09-05 (Estimated); Study Completion 2021-10-05 (Estimated)

PRIMARY OUTCOMES:
1. numerical rating pain score (NRS) during the course of delivery | every 30 minutes throughout the delivery
  1. numerical rating pain score (NRS) during the course of delivery will be recorded and compared

SECONDARY OUTCOMES:
1. the total doses of pethidine needed through-out delivery will be measured | throughout the first stage of delivery
2. the incidence of failed delivery and need of cesarean section will be assessed | throughout delivery time
3. the incidence of transient fetal bradycardia or deceleration after the administration of the block will be recorded | immediately after administration of the block
4. ABGAR score of the neonate immediately after delivery and after 5min, 10min,15min after delivery. Will be recorded | at birth , after 5 min., 10min., 15 min.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt